CLINICAL TRIAL: NCT06169774
Title: Video Training Supplementation to Reduce the Risk of Central Venous Catheter Infection in Patients Discharged on Home Parental Nutrition
Brief Title: Video Training Supplementation for Patients Discharged on Home Parental Nutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB23-1285
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Intestinal Failure
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video (Experimental): Participants will be asked to watch an education video addressing aseptic techniques to safely handle central catheters at home during parenteral nutrition infusions.
  Interventions: Other: Educational video
- No educational video (No Intervention): Participants will be managed according to routine care.

INTERVENTIONS:
Other: Educational video — Watch the 17-minute educational video as many times as needed within a 12-month period.
  Arms: Educational video

SUMMARY:
The goal of this clinical trial is to develop an educational video addressing the aseptic techniques to safely handle central catheters for administrating parenteral nutrition at home.

DETAILED DESCRIPTION:
Home parenteral nutrition is an alternative form of providing nutrition to people whose digestive systems either can't absorb or tolerate food eaten by mouth. Parenteral nutrition provides liquid nutrients, including carbohydrates, proteins, fats, vitamins, minerals and electrolytes. In recent years, more emphasis has been placed on delivering parenteral nutrition to patients at home. Studies have shown that patients receiving home parenteral nutrition are at higher risk for bloodstream infections compared to other patients with chronic infusion needs. Catheter-related bloodstream infection is a major cause of mortality and morbidity in patients receiving parenteral nutrition. It is important to maintain safe vascular access to prevent life-threatening complications. This study aims to assess the effectiveness of the video training on the rate of catheter related bloodstream infection over a 12-month period of time.

ELIGIBILITY:
Inclusion Criteria:

* Taking home parenteral nutrition for the first time
* Willing to self-administer parenteral nutrition
* Age ≥ 18 yrs
* Able to provide informed consent
* Able speak and understand English

Exclusion Criteria:

* Already taking home parenteral nutrition
* not willing to self-administer parenteral nutrition
* Age < 18 years-old
* Unable to provide informed consent
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis of catheter related bloodstream infection (CRBI) events | baseline-12 months
  Change in number of CRBI events measured by complete blood count test.

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Micic, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT06169774/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT06169774/ICF_001.pdf